CLINICAL TRIAL: NCT03562819
Title: An Observational, Multicentre, Prospective Study to Evaluate Concordance of Detecting EGFR (Epidermal Growth Factor Receptor) Mutation by Circulating Tumour Free DNA Versus Tissues Biopsy in NSCLC (Non-small Cell Lung Cancer).
Brief Title: Study to Evaluate Concordance of Detecting EGFR (Epidermal Growth Factor Receptor) Mutation by Circulating Tumour Free DNA Versus Tissues Biopsy in NSCLC (Non-small Cell Lung Cancer).
Acronym: CONCORDANCE
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D5161R00003
Record Dates: First submitted 2018-05-22; First posted 2018-06-20 (Actual); Last update posted 2020-06-05 (Actual); Status verified 2020-06

CONDITIONS: NSCLC (Non-small Cell Lung Cancer)
Keywords: Epidermal Growth Factor Receptor
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- NSCLC: Non-small cell lung cancer

SUMMARY:
This is a multicentre, prospective, study of EGFR )Epidermal Growth Factor Receptor) mutation status in advanced NSCLC (Non-small cell lung cancer)patients (locally advanced and/or metastatic disease) with adenocarcinoma histology proposed to be conducted at 15 sites from different geographical regions across India. The study targets to enrol 268 patients over a period of 6 months.

DETAILED DESCRIPTION:
This is a multicentre, prospective, study of EGFR mutation status in advanced NSCLC patients (locally advanced and/or metastatic disease) with adenocarcinoma histology proposed to be conducted at 15 sites from different geographical regions across India. The study targets to enrol 268 patients over a period of 6 months. The study will enroll patients with histologically confirmed, systemic treatment naïve adenocarcinoma metastatic cancer (stage IV). This will be a single visit study. No study medication will be prescribed or administered as a part of study procedure.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who provide written informed consent
2. Patients aged 18 years and older
3. Newly diagnosed patients with Metastatic (stage IV) NSCLC.
4. Histologically confirmed Adenocarcinoma NSCLC patient as per tissue biopsy and Tissue sample sent for EGFR mutation analysis OR result for EGFR mutation test is available from last 28 days from the date of enrolment.
5. Patient should be naïve for any systemic treatment (i.e. no chemotherapy or EGFR-TKI)

Exclusion Criteria:

1. Patient with any medical condition that, in the opinion of the investigator, would interfere with outcome of the study
2. Patient participating in any other interventional clinical study/trial.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: NSCLC (Non-small cell lung cancer)
Sampling Method: Probability Sample
Enrollment: 268 (Actual)
Dates: Start 2018-08-16 (Actual); Primary Completion 2019-06-07 (Actual); Study Completion 2019-06-07 (Actual)

PRIMARY OUTCOMES:
Determine the level of concordance between EGFR mutation status | 1 Day
  by tissue and plasma based testing in terms of Overall Concordance, Sensitivity, specificity, Positive predictive value & negative predictive value.

SECONDARY OUTCOMES:
Assess the frequency of T790M mutation among study patients. | 1 Day
  Frequency and percentage of TKI treatment naïve NSCLC patients with T790M mutation will be provided.

CONTACTS AND LOCATIONS:
Locations (10):
- India (10):
  - Reserch Site, Punjab, Chandigarh
  - Research Site, Bengaluru, Karnataka
  - Research Site, Kerala, Kozhikode
  - Research Site, Mumbai, Maharashtra
  - Research Site, Maharashtra, Mumbai
  - Research Site, New Delhi, National Capital Territory of Delhi
  - Research Site, Bhubaneswar, Odisha
  - Research Site, Hyderabad, Telanagana
  - Research Site, Kolkata, West Bangal
  - Research Site, Kolkata, West Bengal

REFERENCES:
- [Derived] Prabhash K, Biswas B, Khurana S, Batra U, Biswas G, Advani SH, Mohapatra PN, Rajappa S, Sharma A, Patil S, Dattatreya PS, Roy R, Almel S, Goyal G, Warrier N. CONCORDANCE: A real-world evidence study to evaluate the concordance of detecting epidermal growth factor receptor (EGFR) mutation by circulating tumor DNA* versus tissue biopsy in patients with metastatic non-small cell lung cancer. Indian J Cancer. 2022 Mar;59(Supplement):S11-S18. doi: 10.4103/ijc.ijc_438_21. PMID 35343188
- See also: Related Info — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D5161R00003&attachmentIdentifier=dfb6fc8b-84d3-4b83-87af-01a058f7a79e&fileName=Concordance_CSR_V1.0_25Mar2020_Synopsys.pdf&versionIdentifier=